CLINICAL TRIAL: NCT04786002
Title: The Therapeutic Window of Busulfan in Children With Haemopoietic Stem Cell Transplantation：A Multicenter Study in China
Brief Title: Target Busulfan Exposure in Children With HSCT in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Children's Hospital of Soochow University (Other); Children's Hospital of Fudan University (Other); Fujian Medical University Union Hospital (Other); Guangzhou Women and Children's Medical Center (Other); West China Second University Hospital (Other); Beijing Children's Hospital (Other); Shenzhen Children's Hospital (Other Government); The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-KY-BXA-01
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: HSCT; busulfan; PPK; EFS
MeSH Terms: interventions — Busulfan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The genetic variants were determined at the following loci: GSTA1-69C/T (rs3957357); -52G/A(rs3957356); -513A/G (rs11964968); -631T/G (rs4715333); -1142C/G(rs58912740) and GSTP1 313A/G (rs1695). Homozygous deletion of the GSTM1 and GSTT1 genes was also determined.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Busulfan — The BU administration regimen was four times a day (Q6h), continuous intravenous infusion for 2 hours, 3 or 4 days in a row.

SUMMARY:
Objectives To evaluate the correlation between BU exposure and post-transplant clinical results (efficacy and safety) to establish the optimal BU treatment window for myeloablative conditioning in Chinese pediatrics, provide theoretical basis and the new strategy for BU individualized dosage, further optimize transplant treatment and reduce drug-related toxicity.

Population 500 participants of any sex between the age of 0.1 and 18 years. Patients receiving the BU-based myeloablative conditioning before transplantation.

Endpoint primary To establish BU pop-PK model and analyze the association between BU AUC and event-free survival (EFS)or overall survival (OS) after transplantation in Chinese pediatrics.

Secondary The investigators are also interested in transplantation-related mortality (TRM), acute toxicity and chronic GvHD.

DETAILED DESCRIPTION:
Objectives To evaluate the influence factors of BU metabolism in children and the correlation between BU exposure and post-transplant clinical results (efficacy and safety) to establish the optimal BU treatment window for myeloablative conditioning in Chinese pediatrics, provide theoretical basis and the new strategy for BU individualized dosage, further optimize transplant treatment and reduce drug-related toxicity.

Endpoint primary The main study endpoints are event-free survival (EFS) and overall survival (OS). EFS is calculated from the time of transplant until death, relapse of disease, or graft failure (defined as non-engraftment or rejection), whichever occurred first. OS is the time between transplantation and death of any cause. All surviving patients are censored at day of last contact. Duration of follow-up is the time from transplant to the last assessment for surviving patients or death.

Secondary The investigators are also interested in transplantation-related mortality (TRM), acute toxicity and chronic GvHD. TRM is defined as death unrelated to underlying disease. Acute toxicities are defined as VOD (diagnosed according to modified Seattle criteria), acute GvHD grade II-IV (diagnosed and graded according to Mount Sinai Acute GvHD International Consortium (MAGIC) criteria, oral mucositis (grade II-IV) and hemorrhagic cystitis (grade II-IV). Two of the most commonly utilised scales for oral mucositis are the WHO and NCI-CTCAE scales. Chronic GvHD should be graded as mild, moderate or severe according to the National Institutes of Health (NIH) consensus criteria.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects or their legal guardians voluntarily sign the informed consent, and can complete the study in accordance with the requirements of the program;
2. No age or gender restriction;
3. Patients with blood disease confirmed by histopathology or cytology;
4. BU-based regimen will be adopted. The BU administration regimen was four times a day (Q6h), continuous intravenous infusion for 2 hours, 3 or 4 days in a row.

Exclusion Criteria:

1. Patients with difficulty in vein blood sampling (if there is a needle, blood history);
2. BU TDM was not performed during the treatment;
3. Subjects who are considered unfit to participate in the trail by the investigator.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 500 participants of any sex between the age of 0.1 and 18 years. Patients receiving the BU-based myeloablative conditioning before transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
event-free survival (EFS) | 2 years after administration of busulfan
  EFS is calculated from the time of transplant until death, relapse of disease, or graft failure (defined as non-engraftment or rejection), whichever occurred first.
overall survival (OS) | 2 years after administration of busulfan
  OS is the time between transplantation and death of any cause.

SECONDARY OUTCOMES:
transplantation-related mortality (TRM) | 2 years after administration of busulfan
  TRM is defined as death unrelated to underlying disease.
acute toxicity | 2 years after administration of busulfan
  Acute toxicities are defined as VOD (diagnosed according to modified Seattle criteria),, acute GvHD grade II-IV (diagnosed and graded according to Mount Sinai Acute GvHD International Consortium (MAGIC) criteria, oral mucositis (grade II-IV) and hemorrhagic cystitis (grade II-IV). Two of the most commonly utilised scales for oral mucositis are the WHO and NCI-CTCAE scales.
chronic GvHD | 2 years after administration of busulfan
  Chronic GvHD should be graded as mild, moderate or severe according to the National Institutes of Health (NIH) consensus criteria

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miao, PhD, Principal Investigator — The First Affiliated Hospital of Soochow University; Shaoyan Hu, MD, Principal Investigator — Children's Hospital of Soochow University
Locations (1):
- the First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

REFERENCES:
- [Background] Dix SP, Wingard JR, Mullins RE, Jerkunica I, Davidson TG, Gilmore CE, York RC, Lin LS, Devine SM, Geller RB, Heffner LT, Hillyer CD, Holland HK, Winton EF, Saral R. Association of busulfan area under the curve with veno-occlusive disease following BMT. Bone Marrow Transplant. 1996 Feb;17(2):225-30. PMID 8640171
- [Background] Bartelink IH, Bredius RG, Belitser SV, Suttorp MM, Bierings M, Knibbe CA, Egeler M, Lankester AC, Egberts AC, Zwaveling J, Boelens JJ. Association between busulfan exposure and outcome in children receiving intravenous busulfan before hematologic stem cell transplantation. Biol Blood Marrow Transplant. 2009 Feb;15(2):231-41. doi: 10.1016/j.bbmt.2008.11.022. PMID 19167683
- [Background] Palmer J, McCune JS, Perales MA, Marks D, Bubalo J, Mohty M, Wingard JR, Paci A, Hassan M, Bredeson C, Pidala J, Shah N, Shaughnessy P, Majhail N, Schriber J, Savani BN, Carpenter PA. Personalizing Busulfan-Based Conditioning: Considerations from the American Society for Blood and Marrow Transplantation Practice Guidelines Committee. Biol Blood Marrow Transplant. 2016 Nov;22(11):1915-1925. doi: 10.1016/j.bbmt.2016.07.013. Epub 2016 Jul 29. PMID 27481448
- [Background] Bartelink IH, Lalmohamed A, van Reij EM, Dvorak CC, Savic RM, Zwaveling J, Bredius RG, Egberts AC, Bierings M, Kletzel M, Shaw PJ, Nath CE, Hempel G, Ansari M, Krajinovic M, Theoret Y, Duval M, Keizer RJ, Bittencourt H, Hassan M, Gungor T, Wynn RF, Veys P, Cuvelier GD, Marktel S, Chiesa R, Cowan MJ, Slatter MA, Stricherz MK, Jennissen C, Long-Boyle JR, Boelens JJ. Association of busulfan exposure with survival and toxicity after haemopoietic cell transplantation in children and young adults: a multicentre, retrospective cohort analysis. Lancet Haematol. 2016 Nov;3(11):e526-e536. doi: 10.1016/S2352-3026(16)30114-4. Epub 2016 Oct 13. PMID 27746112
- [Background] Ansari M, Theoret Y, Rezgui MA, Peters C, Mezziani S, Desjean C, Vachon MF, Champagne MA, Duval M, Krajinovic M, Bittencourt H; Pediatric Disease Working Parties of the European Blood and Marrow Transplant Group. Association between busulfan exposure and outcome in children receiving intravenous busulfan before hematopoietic stem cell transplantation. Ther Drug Monit. 2014 Feb;36(1):93-9. doi: 10.1097/FTD.0b013e3182a04fc7. PMID 24061446
- [Background] Nava T, Kassir N, Rezgui MA, Uppugunduri CRS, Huezo-Diaz Curtis P, Duval M, Theoret Y, Daudt LE, Litalien C, Ansari M, Krajinovic M, Bittencourt H. Incorporation of GSTA1 genetic variations into a population pharmacokinetic model for IV busulfan in paediatric hematopoietic stem cell transplantation. Br J Clin Pharmacol. 2018 Jul;84(7):1494-1504. doi: 10.1111/bcp.13566. Epub 2018 Apr 27. PMID 29469189